CLINICAL TRIAL: NCT00434928
Title: Dietary Intake and Nutrient Status of Children With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Dietary Intake and Nutrient Status of Children With ADHD
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Eli Lilly and Company (Industry)
Other Study IDs: H05-70464; W05-0185
Record Dates: First submitted 2007-02-13; First posted 2007-02-14 (Estimated); Last update posted 2007-02-14 (Estimated); Status verified 2007-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: observational; dietary intake; nutrient status; serum assessors; Attention-Deficit/Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Assess the dietary intake of children aged 6-12 years by means of a 24-hour recall and 3-day food record and asses the nutrient status of Vitamin B6, serum ferritin, serum zinc and serum copper of the same children by means of standard laboratory assessments.

DETAILED DESCRIPTION:
* To document the use of vitamin and vitamin-mineral supplements
* To determine the percent consumption of low nutrient density (LND) foods
* To compare the dietary intake of ADHD children with the established standards of the Dietary Reference Intakes (DRIs)
* To compare the dietary intake of children with ADHD to the dietary recommendations of Canada's Food Guide for Healthy Eating
* To determine whether dietary intake is moderated by drug treatment
* To assess the pyridoxal-5'-phosphate (PLP), serum ferritin, serum zinc, and serum copper status of ADHD by standard laboratory blood test
* to measure height and weight in ADHD children

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of ADHD
* Age 6-12 years inclusive

Exclusion Criteria:

* No use of medication that affects dietary intake (eg. Risperdal)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60
Dates: Start 2006-01; Study Completion 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Margaret D. Weiss, MD, Principal Investigator — University of British Columbia
Locations (1):
- Provincial ADHD Program, BC Children's Hospital, Vancouver, British Columbia, Canada